CLINICAL TRIAL: NCT01273844
Title: Study of the Combination of Bortezomib and Dexamethasone Followed by HSCT in AL
Brief Title: Study of Bortezomib +HSCT in Primary Systemic Amyloidosis (AL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-Hong Liu, M.D. (Other)
Collaborators: Soochow University (Other); Nanjing Medical University (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1006
Record Dates: First submitted 2011-01-03; First posted 2011-01-11 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Amyloidosis
Keywords: hematopoietic stem cell transplantation; amyloidosis; Bortezomib
MeSH Terms: conditions — Amyloidosis | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): Patients will receive two 21-day cycles of induction therapy with vel / dex regimen. Bortezomib 1.3mg/m2 on days 1, 4, 8 and 11 will be given by intravenous bolus injection while Dexamethasone 40 mg/d will be taken orally on days 1-4.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib
  Other Names: autologous hematopoietic stem cell transplantation

SUMMARY:
To evaluate the efficacy and safety of Vel-Dex therapy (bortezomib and dexamethasone) followed by autologous hematopoietic stem cell transplantation as an initial treatment in patients with newly diagnosed AL.

DETAILED DESCRIPTION:
Patients will receive two 21-day cycles of induction therapy with vel / dex regimen. Bortezomib 1.3mg/m2 on days 1, 4, 8 and 11 will be given by intravenous bolus injection while Dexamethasone 40 mg/d will be taken orally on days 1-4. After two cycles of vel / dex therapy, the collection of peripheral blood stem cells (PBSC) should be completed within 4 weeks.Patients will receive ASCT therapy in 8 weeks after collection of PBSC (Recorded as day 0), while melphalan (day -2) with a dose of 100,140 or 200 mg/m2 (choosing a dose according to the degree of risk for patients ) and Vel 1mg/m2 (days -6, -3, +1, +4) will be given. Four additional 21-day cycles of Vel treatment (with a dose of 1.6mg/m2 on day 1 and 8 of the cycle) will be conducted as consolidation therapy during the recommended 60-90 days after HSCT, or after resumption of hematopoietic function ( neutrophil count > 1.5x109/L and platelet count> 50x109/L). Later patients won't need maintenance therapy.

The efficacy criteria are the international standards set with consensus of experts in the Tenth International Symposium on Amyloid and Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. aged 18-65 years;
3. Patients with newly diagnosed AL;
4. Appropriate for autologous hematopoietic stem cell transplantation;
5. Abnormal M protein or free light chain detected in serum and / or urine
6. ECOG score 0-2 points;
7. Subjects (or their legal representatives) must signed an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.

Exclusion Criteria:

1. Subjects received systematic treatment with steroids
2. Subjects received plasmapheresis to treat clinical significant hyperviscosity syndrome within 4 weeks before enrollment.
3. Pregnant and breastfeeding women;
4. Subjects suffering from multiple myeloma.
5. hypersensitivity to dexamethasone, bortezomib, mannitol, boron, or heparin (if use catheters);
6. Subjects have severe cardiovascular disease,
7. Subjects have serious physical disease and mental illnesses which may interfere the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 12 months
  Complete response rate at 12 months post-transplantation

SECONDARY OUTCOMES:
overall response rate | 12 months
  overall response rate(ie.,CR + PR) at 12 months post-transplantation

OTHER OUTCOMES:
progression-free survival | 2 years
  progression-free survival (PFS) at 2 years post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: zhihong Liu, Master, Principal Investigator — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, China
Locations (1):
- Soochow University, Suzhou, Jiangsu, China